CLINICAL TRIAL: NCT07214831
Title: A Feasibility and Acceptability Study of a Large Language Model-based Conversational Agent for Brief Alcohol Intervention Among Emerging Adults
Brief Title: A Feasibility and Acceptability Study of a Large Language Model-based Chatbot for Brief Alcohol Intervention Among Emerging Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Russell, Alex, Assistant Professor of Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P001459; R34AA032472 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Large language model-based chatbot brief alcohol intervention (Experimental): All participants will interact with a large language model-based chatbot designed to deliver a brief alcohol intervention session.
  Interventions: Behavioral: Large language model-based chatbot brief alcohol intervention session

INTERVENTIONS:
Behavioral: Large language model-based chatbot brief alcohol intervention session — The intervention is a large language model-based chatbot designed to delivered brief alcohol interventions using motivational interviewing-consistent strategies. The chatbot session will last approximately 45 minutes and will include a decisional balance exercise, feedback on drinking patterns, normative beliefs about drinking, alcohol-related consequences, goal setting, and harm-reduction strategies.

SUMMARY:
American emerging adults (EAs; aged 18-29 years) have the highest rates of alcohol use disorder (AUD) and the lowest levels of treatment engagement of any age group. Innovative, scalable, and cost-effective strategies are needed to expand early detection and intervention for EAs engaged in patterns of drinking associated with AUD. Because digital technology use is frequent among EAs, digital interventions may be a particularly suitable way to reach this population. Prior studies of digital alcohol interventions demonstrate modest but consistent reductions in alcohol use, but these tools are often limited by a lack of interactivity and personalization. Large language model (LLM)-based chatbots, such as ChatGPT, may address these limitations by enabling personalized, adaptive, and human-like engagement. These features have the potential to increase uptake and engagement with screening and brief interventions among EAs. This study will develop, validate, and conduct an open trial of an LLM-based chatbot-delivered brief intervention designed to reduce alcohol use and problems among EAs, with the primary goal of establishing preliminary feasibility and acceptability.

DETAILED DESCRIPTION:
This feasibility and acceptability study will develop, validate, and conduct a Phase I single-arm open trial of a large language model (LLM)-based chatbot-delivered brief intervention designed to reduce alcohol use and problems among EAs. To develop the augmented LLM, the investigators will use instruction fine-tuning to enhance conversational abilities within the context of brief interventions based on high-fidelity recordings of sessions from prior clinical trials and simulated patient-provider interactions. A retrieval augmented generation system will be developed to ensure the model delivers accurate information. The augmented LLM will be incorporated into a chatbot interface delivered through a user-friendly web application. To validate the chatbot's capability for delivering brief alcohol interventions, patient actors (clinical or counseling psychology PhD students) will be assigned clinical vignettes depicting diverse EAs with patterns of drinking associated with alcohol use disorder. Patient actors will engage in two randomly ordered online text-based brief intervention sessions for each vignette (one with the chatbot and one with a human clinician). Blinded transcripts from sessions will be reviewed by experts to assess treatment fidelity. To maximize and test initial feasibility and acceptability of the intervention, the investigators will conduct semi-structured interviews with 20 EAs who report hazardous drinking, followed by an open trial with another 20 EAs.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years old
* Engaged in past-month hazardous drinking (consuming ≥ 5/4 drinks for men/women on two or more occasions in the past month) or exceeded recommended guidelines for risky drinking (> 14/7 drinks per week for men/women)
* Able to read and comprehend English at a 5th grade level

Exclusion Criteria:

* Report a history of or active psychosis
* Previous or current engagement in alcohol or drug treatment
* Risk for alcohol withdrawal as evidenced by very heavy weekly drinking reports on the alcohol screener (> 40 standard drinks in a typical week in the past month)
* Demonstrate inability or unwillingness to attend in-person office visits
* Demonstrate inability or unwillingness to identify an emergency contact who could be contacted in case the participant becomes lost to follow-up

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2027-06-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to achieve target enrollment | Enrollment
  Recruitment feasibility will be evaluated based on the length of time needed to recruit target enrollment (N = 20)
Rate of participant retention | 1-month post intervention1-month post intervention
  Retention feasibility will be achieved if >80% of participants who consented to participating in the study complete one-month follow-up assessment.
Acceptability (System Usability Scale) | Immediate post-intervention session
  Acceptability of the conversational agent-delivered intervention will be measured using the 10-item System Usability Scale. Each question is rated on a Likert-type scale ranging from (1) strongly disagree to (5) strongly agree.
Acceptability - intervention delivery method | Immediate post-intervention session
  Percentage of participants who agree or strongly agree the intervention delivery method was acceptable
Acceptability - usable | Immediate post-intervention session
  Percentage of participants who agree or strongly agree the intervention was easy to interact with
Acceptability - helpful | Immediate post-intervention session
  Percentage of participants who agree or strongly agree the intervention was helpful
Acceptability - recommend to others | Immediate post-intervention session
  Percentage of participants who agree or strongly agree they would recommend the chatbot to others

SECONDARY OUTCOMES:
Motivation to change drinking (Readiness Ruler) | Enrollment, immediate post-intervention session, and 1 month post-intervention
  Motivation to change drinking will measured using the Readiness Ruler.
Daily drinking questionnaire (DDQ) | Enrollment and 1 month post-intervention
  Past-month typical drinks per week and frequency of heavy drinking will be assessed using the DDQ. Respondents are asked to record the number of drinks they consume each day of a typical week over the previous month.
Alcohol Use Disorders Identification Test (AUDIT) | Enrollment and 1 month post-intervention
  Past-month frequency of heavy drinking will be assessed using the AUDIT, a 10-item screening tool used to identify hazardous and harmful drinking patterns. Total scores range from 0 to 40, with higher scores indicating more hazardous or harmful drinking patterns.
Young Adult Alcohol Consequences Questionnaire (YAACQ) | Enrollment and 1 month post-intervention
  Alcohol-related problems will be assessed using the YAACQ. Respondents will be asked to indicate (yes/no) which of the 48 potential problems they have experienced as a result of their drinking over the previous month.
Protective behavioral strategies scale (PBSS) | Enrollment and 1 month post-intervention
  Protective behavioral strategies will be assessed using the 15-item PBSS. Participants will be asked to indicate how often they used each strategy when drinking alcohol during the previous month. Response options are presented on a 6-point Likert type scale ranging from 1 (never) to 6 (always).
Alcohol treatment utilization | Enrollment and 1 month post-intervention
  Alcohol treatment utilization, including a variety of options, will be measured by asking respondents to indicate (yes/no) which of the potential options they have utilized.

CONTACTS AND LOCATIONS:
Overall Officials: Alex M Russell, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be submitted to the NIAAA Data Archive in accordance with NIH requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: De-identified individual participant data (IPD) and supporting documents will be deposited in the NIAAA Data Archive (NIAAADA) hosted within the NIMH Data Archive. Data will be submitted within 6 months of collection and will be available after study completion, in perpetuity.
Access Criteria: Data will be de-identified and available as public use data through the NIAAA Data Archive. Access requires submission of a data use request through the NIAAADA and agreement to the Terms of Use, which limit use to scientific research, prohibit attempts to identify participants, and require reporting of any breaches of confidentiality.
URL: https://nda.nih.gov/